CLINICAL TRIAL: NCT07255391
Title: Application of Platelet-rich Plasma for Healing og Grade III Ulcer.
Brief Title: Use of PRP for the Healing of Grade III Ulcers
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssaigPRPBE0205; BE0205 (Other: Fundació per la Recerca Mutua Terrassa)
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: PRP Injection; Ulcer
Keywords: PRP; Úlceras Grado III
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Intervention Model Description: Control y experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Group receiving treatment with PRP
  Interventions: Procedure: PRP group
- Control Group (Active Comparator): Group receiving standard/traditional care
  Interventions: Procedure: Classic treatment

INTERVENTIONS:
Procedure: PRP group — The PRP will be injected into the wound bed, unlike in other studies where it has been used only as a gel.
  Arms: Experimental Group
Procedure: Classic treatment — Standard care for patients in the control group: Aquacel + Gel every 48 hours
  Arms: Control Group

SUMMARY:
Treatment with platelet-rich plasma (PRP) consists of extracting a small amount of blood from the patient himself, which is later processed by centrifugation to obtain a fraction rich in platelets. It will be done on weekly or fortnightly blood extraction procedure, depending on the process. Between 1-3 sterile citrate collection tubes will be used, which may vary depending on the size of the ulcer. Each tube can contain approximately 8-10ml of blood and the procedure is carried out under aseptic conditions and with material from a single use Once the sample has been centrifuged, the blood plasma will be extracted and the concentrate obtained will be applied directly on the wound or ulcer with the objective of stimulating and accelerating healing by means of growth factors.

This procedure is used as complementary therapy in chronic ulcers or with difficulty in healing, such as they can be venous, arterial, pressure or diabetic foot ulcers.

DETAILED DESCRIPTION:
1. Introduction

   Platelet-rich plasma (PRP) is an autologous blood derivative obtained by centrifuging the patient's own blood. It contains a high concentration of growth factors that promote tissue regeneration and cell proliferation. Its use in the treatment of chronic ulcers has shown good results, especially in wounds that do not respond to conventional treatments.
2. Required Materials

   Sterile 5 ml and 10 ml syringes

   Needles or butterfly needle and 20G vacutainer for extraction, and 30G (4 mm or 13 mm) for infiltration

   Tube with anticoagulant (3.8% sodium citrate), closed system technique

   Clinical centrifuge with fixed-angle or swinging-bucket rotor

   Gloves, mask, gown, and sterile working surface

   Sterile dressings, saline solution, and antiseptics
3. Blood Extraction

   Draw between 10 and 20 ml of venous blood from the patient, depending on the extent of the ulcer. Use tubes with anticoagulant to prevent premature coagulation.

   Apply a closed system technique to avoid handling and contamination of the sample.
4. Centrifugation

   Use a single centrifugation cycle to obtain high-quality PRP: 3500 rpm for 10 minutes.

   Once the process is complete, prepare the PRP in the selected 5 ml or 10 ml syringes.
5. PRP Application

   → Before application:

   Clean the wound with saline solution and antiseptic.

   Perform debridement if there is necrotic or fibrinous tissue.

   → Application methods:

   Intradermal or subdermal perilesional infiltration using a fine needle (30G 4 mm or 30G 13 mm).

   Direct application of PRP onto the wound bed.

   Apply a topical layer.

   Cover with a sterile dressing or gauze soaked in the same PRP.
6. Monitoring and Follow-Up

   Evaluate the wound weekly or biweekly.

   Repeat treatment every 1-2 weeks depending on progress.

   Take photographs and document each visit to assess clinical response.
7. Contraindications and Precautions

   Severe thrombocytopenia (< 100,000 platelets/μL)

   Active systemic infection

   Severe hematological disorders

   Do not administer in case of allergy to the anticoagulants used

   Active local infection
8. Conclusions

PRP represents an innovative and safe therapeutic option in the management of chronic ulcers, with good clinical outcomes and minimal side effects when performed using the appropriate technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Grade III ulcers.
* Patients with ulcers older than two weeks.
* Patients with an optimal platelet count according to prior laboratory tests.

Exclusion Criteria:

* Patients with a palliative profile.
* Patients with a limited life expectancy.
* Patients with a platelet count below 10 × 10⁹/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in ulcer diameter at 30, 60, and 90 days | At the beginning of patient inclusion and at 30, 60, and 90 days from the start of therapy

SECONDARY OUTCOMES:
Scoring on the PUSH Scale | At the beginning of the study, and at 30, 60, and 90 days from the start of the therapy
  The PUSH Scale assesses the area of the pressure ulcer (scored from 0 to 10), the amount of exudate (scored from 0 to 3), and the type of tissue (scored from 0 to 4). The higher the total score, the worse the condition of the ulcer
Amount of Exudate | At the time of patient inclusion, and at 30, 60, and 92 days from the start of treatment
  Amount of ulcer exudate, scored from 0 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Atenció Intermitja l'Ametlla del Vallès, L'Ametlla del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All patient data will be stored in the REDCAP system, which ensures the protection of patients' personal data.
Supporting Information: SAP
Time Frame: he data will be accessible only to the principal investigators of the study, from the start of the study (November 2025) until the completion of the data analysis (February 2028)
Access Criteria: Only the principal investigators of the study will have access to the data, and the data can only be accessed through the REDCAP application

REFERENCES:
- [Background] Sánchez-García S, Fernández-Parra R, Villanueva E, García-Hernández A, García-García F, García-Sánchez E. Uso del plasma rico en plaquetas en el tratamiento de úlceras vasculares: nuestra experiencia. Angiología. 2020;72(1):15-22.
- [Background] Lázaro-Martínez JL, García-Álvarez Y, García-Morales E, Alvaro-Afonso FJ, Molines-Barroso RJ. Eficacia del plasma rico en plaquetas en la cicatrización de úlceras del pie diabético: una revisión sistemática y metaanálisis. Endocrinol Diabetes Nutr. 2019;66(3):187-94.
- [Background] Knighton DR, Doucette M, Fiegel VD, Ciresi K, Butler E, Austin L. The use of platelet derived wound healing formula in human clinical trials. Prog Clin Biol Res. 1988;266:319-29. No abstract available. PMID 3289047
- [Background] Rodriguez-Flores J, Palomar-Gallego MA, Enguita-Valls AB, Rodriguez-Peralto JL, Torres J. Influence of platelet-rich plasma on the histologic characteristics of the autologous fat graft to the upper lip of rabbits. Aesthetic Plast Surg. 2011 Aug;35(4):480-6. doi: 10.1007/s00266-010-9640-5. Epub 2010 Dec 24. PMID 21184066